CLINICAL TRIAL: NCT00665678
Title: Neural Correlates of Early Intervention for PTSD
Brief Title: Neural Correlates of Early Intervention for Posttraumatic Stress Disorder (PTSD)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Foundation for Atlanta Veterans Education and Research, Inc. (Other)
Collaborators: Emory University (Other)
Responsible Party: James Douglas Bremner, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDMRP PT074585
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): paroxetine
  Interventions: Drug: paroxetine
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: paroxetine — treatment for three months with paroxetine
  Arms: 1
Drug: placebo — treatment for three months with placebo
  Arms: 2

SUMMARY:
Background: Innovation: Over 150,000 soldiers are currently deployed in Iraq as part of Operation Iraqi Freedom (OIF), and 12% of returning OIF veterans have posttraumatic stress disorder (PTSD). Research from our group and others showed lasting neurobiological consequences of PTSD, including increased amygdala function and decreased medial prefrontal function, verbal declarative memory problems, and smaller hippocampal volume that reverses with treatment with the serotonin reuptake inhibitor (SSRI) paroxetine or the anticonvulsant phenytoin. Recently we found that three months of treatment with paroxetine in PTSD patients resulted in an increase in hippocampal N-acetyl-aspartate (NAA), a marker of neuronal integrity, as well as decreased brain metabolism in the amygdala and a reversal or stress induced decreases in medial prefrontal function. Subjects treated with placebo did not have an increase in NAA, however subsequent treatment for three months with open label paroxetine resulted in an increase in NAA to the level seen in the subjects treated with paroxetine in the double-blind phase. Paroxetine was associated with a decrease in amygdala metabolism measured with positron emission tomography (PET) and increased medial prefrontal function. Intervening soon after the trauma is critical for long-term outcomes, since with time traumatic memories become indelible and resistant to treatment. Diminished efficacy of treatment over time is shown by the fact that trials of Vietnam veterans have shown less efficacy over the years. Animal studies show that pretreatment before stress with antidepressants reduces chronic behavioral deficits related to stress; although for ethical and other reasons no studies have provided pretreatment before trauma exposure in humans. In our current VA Merit funded program we are looking at the effects of early interventions for Iraq soldiers with paroxetine, looking at chronicity of PTSD, cognition, cortisol response to stress, hippocampal volume and NAA, as outcomes. We now propose to add measurement of neural correlates of paroxetine response using PET.

Objectives/Hypotheses: The objectives of this research are to:

* Assess the efficacy of paroxetine versus placebo in the treatment of early PTSD in OIF veterans
* Assess the effects of paroxetine versus placebo on amygdala metabolism and medial prefrontal response to stress in OIF veterans with PTSD.
* Assess the ability of brain imaging to predict treatment response and to identify veterans with early PTSD who will benefit from early interventions.

Hypotheses are that paroxetine will be associated with: 1) an improvement in PTSD symptoms compared to placebo based on the change in the CAPS from baseline to three months of treatment in veterans of OIF; 2) increased medial prefrontal function and decreased amygdala metabolism in veterans of OIF.

Specific Aims:

* Compare paroxetine to placebo in the treatment of early PTSD in OIF veterans
* Measure amygdala metabolism and medial prefrontal response to stress with PET in OIF veterans with PTSD before and after paroxetine or placebo treatment.

DETAILED DESCRIPTION:
Study Design: Subjects returning from Iraq who meet criteria for early PTSD (N=160) will be included in the study with a recruitment goal of 144 completers. A group of 80 healthy subjects with a history of military service during the period of OIF without a history of deployment and without PTSD and 80 healthy subjects with a history of deployment without PTSD will serve as comparator groups. All subjects will undergo baseline imaging of the brain with PET FDG and with measurement of brain blood flow during a memory task and with exposure to trauma related reminders (slides and sounds) and MRI and baseline psychometric assessments, following which PTSD subjects will be randomized to receive paroxetine or placebo for three months, with repeat imaging and assessments. After this PTSD subjects will be treated with three months of open label paroxetine, followed by a repeat of imaging and assessments. This will be an intent to treat analysis, therefore all subjects who were randomized and took at least one dose of study medication will be assessed at three months, regardless of whether they were able to stay on study medication. This will complement our currently VA Clinical Trial Merit funded application to measure hippocampal volume, NAA, and cortisol response to stress before and after early intervention with paroxetine in returning Iraq vets with early PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Male and female veterans age 18-50
* Returned from Iraq Theater within the past six months
* Screen positive for PTSD related to Iraq deployment based on the PTSD Checklist
* Confirmed with PTSD based on the CAPS, including one month duration of symptoms
* Being discharged from active service from Iraq
* Provide written informed consent

Exclusion Criteria:

* History of loss of consciousness of more than one minute
* Psychotropic medication use within the previous four weeks
* History (based on the SCID) of lifetime or current alcohol or substance abuse/dependence, schizophrenia, schizoaffective disorder, or bipolar disorder.
* Positive urine toxicology screen
* History of pre-deployment-related PTSD or partial PTSD based on the CAPS
* History of PTSD or partial PTSD related to a prior deployment
* Serious medical or neurological illness
* Pregnancy
* History of asthma
* Steroid usage, both inhaled and oral
* Seizure disorder
* Prenatal/perinatal substance exposure or trauma.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2008-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
PTSD symptoms as measured with the CAPS | three months

SECONDARY OUTCOMES:
Assess the effects of paroxetine versus placebo on amygdala metabolism and medial prefrontal response to stress in OIF veterans with PTSD. | three months

CONTACTS AND LOCATIONS:
Overall Officials: James D Bremner, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- See also: Dr. Bremner's Home Page — http://www.dougbremner.com